CLINICAL TRIAL: NCT04620889
Title: A Retrospective Patient Registry on the Long-Term Safety and Performance of the LifeSpan® ePTFE Vascular Graft Used in Open Vascular Surgery
Brief Title: LeMaitre LifeSpan® ePTFE Vascular Graft Retrospective Registry
Status: Completed | Type: Observational
Sponsor: LeMaitre Vascular (Industry)
Responsible Party: Sponsor
Other Study IDs: LFP-15-001
Record Dates: First submitted 2020-11-03; First posted 2020-11-09 (Actual); Last update posted 2024-10-18 (Actual); Status verified 2024-10

CONDITIONS: Diseased or Occluded Blood Vessels; Arteriovenous Shunting for Blood Access

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

GROUPS / COHORTS (2):
- PVP (peripheral vascular disease): Bypass or reconstruction of diseased or occluded blood vessels
  Interventions: Device: PVP
- AV Access (arteriovenous access): Arteriovenous shunting for blood access and bypass.
  Interventions: Device: AV Access

INTERVENTIONS:
Device: AV Access — Arteriovenous shunting for blood access.
  Groups: AV Access (arteriovenous access)
Device: PVP — Bypass or reconstruction of diseased or occluded blood vessels
  Groups: PVP (peripheral vascular disease)

SUMMARY:
This is a post-market, single-arm, retrospective registry. The investigator or its representative will identify eligible patients through a medical record search.

DETAILED DESCRIPTION:
This is a post-market, single-arm, retrospective registry. The investigator or its representative will identify eligible patients through a medical record search. Data will be captured retrospectively. Subjects will have been treated with the investigational device in the past and according to standard of care. Subjects will not be involved in any registry related procedures.

ELIGIBILITY:
Inclusion Criteria:

* Subject has undergone surgical treatment with the LifeSpan.
* Surgical treatment was for bypass or reconstruction of diseased or occluded blood vessels (PVP group) or arteriovenous shunting for blood access (AV group).
* For PVP group: Subject's surgical treatment was at minimum 3 years ago, and maximum 10 years ago, at time of enrollment.
* For AV group: Subject's surgical treatment was at minimum 2 years ago, and maximum 10 years ago, at time of enrollment.

Exclusion Criteria:

* None

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: This is a retrospective registry. The included population is therefore directly representative of the population in a real-world environment.
Sampling Method: Non-Probability Sample
Enrollment: 153 (Actual)
Dates: Start 2020-11-27 (Actual); Primary Completion 2023-11-24 (Actual); Study Completion 2023-11-24 (Actual)

PRIMARY OUTCOMES:
Percentage of vessels patent without requiring intervention to remain open | 3 years
  Percentage of patients exempt from thrombosis/ occlusion and/or restenosis of the target lesion during follow-up
Percentage of vessels patent without requiring intervention to remain open | 2 years
  Percentage of patients exempt from thrombosis/ occlusion and/or restenosis of the target lesion during follow-up

SECONDARY OUTCOMES:
Procedure type | Day of procedure
  Type of procedure
Intra-operative technical success | Day of procedure
  Percentage of patients with proper functioning of the device in the opinion of the investigator at time of surgery
Percentage of vessels patent without requiring intervention to remain open at 1 and 5 year primary patency | 1 year and 5 year
  Percentage of patients exempt from thrombosis/ occlusion and/or restenosis of the target lesion during follow-up
Percentage of vessels patent with intervention to remain open at 1 and 5 year | 1 year and 5 year
  Percentage of patients exempt from thrombosis/ occlusion and/or restenosis of the target lesion during follow-up after interventions
Percentage of vessels patent with intervention to remain open at 1 and 5 year for AV Access | 2 year
  Percentage of patients exempt from thrombosis/ occlusion and/or restenosis of the target lesion during follow-up after interventions
Percentage of vessels patent with intervention to remain open at 1 and 5 year for PVP Group | 3 year
  Percentage of patients exempt from thrombosis/ occlusion and/or restenosis of the target lesion during follow-up after interventions

CONTACTS AND LOCATIONS:
Locations (1):
- Klinikum Nordfriesland GmbH, Husum, Germany

IPD SHARING:
Plan to Share IPD: No
This is a fully anonymized registry. No IPD will be collected or shared.